CLINICAL TRIAL: NCT01389895
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Effect of AMG 557 in Subjects With Subacute Cutaneous Lupus Erythematosus
Brief Title: Safety Study of AMG 557 in Subjects With Subacute Cutaneous Lupus Erythematosus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20100037
Record Dates: First submitted 2011-06-23; First posted 2011-07-08 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Cutaneous Lupus; Lupus
Keywords: Lupus; Cutaneous lupus
MeSH Terms: interventions — AMG 557

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 557 (Active Comparator): All will receive AMG 557 on Day 1, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, and Day 99.
  Interventions: Drug: AMG 557
- AMG 557 Placebo (Placebo Comparator): All will receive placebo on Day 1, Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85, and Day 99.
  Interventions: Drug: AMG 557 Placebo

INTERVENTIONS:
Drug: AMG 557 — AMG 557 (210 mg) or (140 mg ) will be administered as subcutaneous injections in the anterior abdomen of the subjects. Twelve subjects will be randomized to receive AMG 557. Beginning on Day 1, subjects will receive either 210 mg AMG 557 or 140 mg AMG 557 once weekly for 3 weeks on Day 1, Day 8, and Day 15 and following with 6 additional doses of AMG 557 every other week on Day 29, Day 43, Day 57, Day 71, Day 85, and Day 99. Subjects will be followed out to Day 253 for safety, efficacy, pharmacokinetic (PK) and pharmacodynamic (PD) assessments.
  Arms: AMG 557
Drug: AMG 557 Placebo — AMG 557 Placebo (210 mg) or (140 mg )will be administered as subcutaneous injections in the anterior abdomen of the subjects. Twelve subjects will be randomized to receive placebo. Beginning on Day 1, subjects will receive placebo once weekly for 3 weeks on Day 1, Day 8, and Day 15 and following with 6 additional doses of placebo every other week on Day 29, Day 43, Day 57, Day 71, Day 85, and Day 99. Subjects will be followed out to Day 253 for safety, efficacy, pharmacokinetic (PK) and pharmacodynamic (PD) assessments.
  Arms: AMG 557 Placebo

SUMMARY:
This study will be a multicenter, randomized, double-blind, placebo-controlled, multiple dose study in which approximately 24 subjects with SCLE will be enrolled. Cohort 1 will consist of 12 subjects (6 AMG 557: 6 placebo) randomized to receive AMG 557 210 mg or matching placebo. Cohort 2 will consist of 12 subjects (6 AMG 557: 6 placebo) randomized to receive AMG 557 140 mg or matching placebo. Enrollment of Cohort 2 (140 mg) will be initiated after enrollment of Cohort 1 (210 mg) is completed.

DETAILED DESCRIPTION:
Cohort 1 will consist of 12 subjects (6 AMG 557: 6 placebo) randomized to receive AMG 557 210 mg or matching placebo. Cohort 2 will consist of 12 subjects (6 AMG 557: 6 placebo) randomized to receive AMG 557 140 mg or matching placebo. Enrollment of Cohort 2 (140 mg) will be initiated after enrollment of Cohort 1 (210 mg) is completed. After Cohort 1 and 2 enrollment has been completed, the emerging PK and PD data will be reviewed to determine if an additional 4-8 subjects with SCLE will be enrolled into the study to address equivocal results from the study. These 4-8 additional subjects will receive the same dose of either 210 mg or 140 mg SC (in an allocation ratio of 1 AMG 557: 1 placebo).

In addition, an open label extension study for participants in this study may be instituted following completion and analysis of results of this study. Initiation of this study will require that an acceptable risk-benefit profile and some evidence of efficacy are observed in the current study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between the ages of 18 and 70 years of age, inclusive, at the time of randomization;
* Body mass index from 18 to 35 kg/m2 at screening;
* Diagnosis of subacute cutaneous lupus erythematosus (SCLE) with or without systemic lupus erythematosus (SLE). SCLE as defined by the Gilliam and Sontheimer classification (J Am Acad Dermatol 1981; 4(4):471-475). SLE is defined by the most recent American College of Rheumatology criteria, including positive antinuclear antibodies (ANA) during screening or by documented history (at least 1:80 by indirect immunofluorescent assay);
* A history of skin biopsy consistent with the diagnosis of SCLE;
* Positive SS-A and/or SS-B antibodies at screening;
* Intolerance of anti-malarial therapy or ≥ 3 months of anti-malarial therapy with residual disease activity as defined by: at least 2 areas with at least level 2 erythema or 3 areas with at least level 1 erythema using cutaneous lupus erythematosus disease area and severity index (CLASI). The total CLASI activity must be ≥ 10;
* Subject must have stable disease activity for 3 months prior to screening in the clinical judgment of the Principal Investigator (PI) with no anticipated changes in therapy;
* Stable dose of topical steroids no stronger than medium-potency (Class III or Class VII) for ≥ 2 weeks from screening is permitted;
* Prednisone ≤ 10 mg/day (or equivalent) is permitted;
* Stable doses of methotrexate ≤ 20 mg/week, azathioprine ≤ 150 mg/day, and 6-mercaptopurine ≤ 150 mg/day for 12 weeks prior to screening are permitted.
* Exclusion Criteria:
* Drug-induced SCLE;
* Any disorder (including psychiatric), condition or clinically significant disease (other than a diagnosis of SCLE, SLE, or Sjögren's syndrome) that would, by its progressive nature and/or severity, interfere with the study evaluation, completion and/or procedures per the investigator's discretion. This includes any age related co-morbidities such as presence of congestive heart failure, angina, chronic obstructive pulmonary disease, and asthma;
* Presence or history of vasculitis (comprising internal organs or extremities or leading to peripheral neuropathy) within the last 3 years, presence or history of active Central Nervous System (CNS) lupus (defined as seizure disorder, cerebral vascular accident, psychosis ascribed to SLE , encephalitis, meningitis, and myelitis) requiring therapy within the last 3 years;
* History of malignancy;
* Signs or symptoms of a viral, bacterial or fungal infection within 30 days of study randomization, or recent history of repeated infections;
* Underlying condition other than SCLE, SLE, Sjögren's syndrome that predisposes one to infections (eg, history of splenectomy);
* Administration of >10 mg/day prednisone (or equivalent) in the 30 days prior to randomization;
* Prior use of any following biological agents: Rituximab, Lymphostat-B, TACl-Ig, and CTLA4-Ig;
* Current treatment (within 3 months or 5 half-lives of screening) with thalidomide, mycophenolate mofetil, cyclosporine, tacrolimus, sirolimus, Intravenous (IV) immunoglobulin, plasmapheresis, oral or IV cyclophosphamide;
* Receiving or has received any investigational drug (or is currently using an investigational device) within the 30 days or 5 half-lives (whichever is longer), prior to receiving the first dose of study medication).
* 29. Use of any other over-the-counter or prescription medications within the 14 days or 5 half-lives (whichever is longer), prior to receiving the first dose of study medication. Acetaminophen (up to 2 g per day) for analgesia and hormone replacement therapy (eg, estrogen, thyroid) will be allowed. In addition, prescription drugs for hypertension or hypercholesterolemia, oral hypoglycemic drugs, or NSAIDs will be allowed; however, NSAIDS are not permitted within 24 hours of skin biopsies to reduce the risk of bleeding. Other medications may be approved following review by the Principal Investigator and the Amgen Medical Monitor. Written documentation of this review and Amgen acknowledgement is required for subject participation;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety evaluation: Subject incidence of treatment-emergent adverse events, vital signs, physical examinations, clinical laboratory safety tests, ECGs, and the incidence of binding and neutralizing antibodies to AMG 557 | 253 Days

SECONDARY OUTCOMES:
Determine the pharmacokinetic (PK) profile of AMG 557 after multiple subcutaneous (SC) doses in subacute cutaneous lupus erythematosus (SCLE) subjects. | 253 Days
Characterize the mean change and variability in serum SS-A and SS-B autoantibodies. | 253 Days
Characterize change in Cutaneous Lupus Erythematosus Disease Area and Severity Index score (CLASI-a) score. | 253 Days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (9):
- United States (6):
  - Research Site, Birmingham, Alabama
  - Research Site, Ann Arbor, Michigan
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Dallas, Texas
- Australia (2):
  - Research Site, Woolloongabba, Queensland
  - Research Site, Carlton, Victoria
- Research Site, Peterborough, Ontario, Canada

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com